CLINICAL TRIAL: NCT03310398
Title: Latent Constructs: Negative-Positive Valence Domains in Anxiety and Depression
Brief Title: Negative-Positive Valence Domains in Anxiety and Depression
Acronym: RDoC
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Martin Paulus, Adjunct Professor of Psychiatry, University of California, San Diego
Other Study IDs: 130554
Record Dates: First submitted 2015-10-23; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood biomarkers: Investigators will assess blood biomarkers including norepinephrine, dopamine, epinephrine, creatinine, soluble cellular adhesion molecules (sICAM, sVCAM), IFN+ (IFN-gamma, IL-6, and TNF-alpha assayed together), and brain-derived neurotrophic factor (BDNF).
  Genetics: Furthermore, as noted later in this section of the application, investigators have identified abnormalities in functioning of key structures (e.g., amygdala and insula) within the brain's anxiety circuitry in anxiety-prone subjects and there is evidence that certain genes (e.g., SLC6A4) influence the extent of activation in these regions. The focus of this project is to determine to what extent variation in CRF system genes (i.e., CRF, CRF-R1, CRF-R2, UCN, UCN2, UCN3) is associated with anxiety disorders.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anxiety: elevated anxiety (as indicated by a GAD-7 score of 8 or higher)
  Interventions: Behavioral: NeuroImaging; Behavioral: Psychophysiological
- Depression: elevated anxiety (as indicated by a GAD-7 score of 8 or higher)
  Interventions: Behavioral: NeuroImaging; Behavioral: Psychophysiological

INTERVENTIONS:
Behavioral: NeuroImaging — standard anatomical and functional imaging
Behavioral: Psychophysiological — Hear rate, Vagal Tone, Skin Conductance, and Startle Reflex Electromyogram

SUMMARY:
Anxiety and depression are highly prevalent and disabling conditions that frequently co-occur, and are costly to the individual and society. Despite important advances in our understanding of these disorders, there is a significant unmet need to identify reliable and clinically useful tests that can predict prognosis, inform treatment choice for a given individual, and improve treatment outcomes. The aim of this project is to fill this critical gap by validating a battery of measures including brain imaging, psychophysiology, behavior, and self-report that will reliably assess positive and negative affect, or valence, system functioning in a broad sample of individuals screened for anxiety and depression as part of their routine primary care visits.

DETAILED DESCRIPTION:
Participants presenting to the UCSD and UCLA primary care clinics will be screened as part of their routine visit using the Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder 7 (GAD-7). Participants who call in will be asked to provide verbal informed consent for phone screening and the IRB approved Screening Questionnaire and the Overall Anxiety Severity and Impairment Scale (OASIS) will be administered.

Participants who remain eligible after the phone screening will be asked to return for a Clinical Interview, Behavioral Session, Biomarker blood draw, (and optional genetics), and Neuroimaging Session.

All participants will be contacted approximately 3-months later and invited to complete the same battery of self-report measures completed during the baseline session (described below). The self-report measures will be administered through a secure on-line survey database. This data will allow investigators to (1) confirm that participants continue to meet initial eligibility criteria and are therefore eligible for the full re-test battery and (2) use baseline measures of positive and negative valence domains to predict changes in symptoms and functioning.

A subset of 50 participants (n=25 from each UCSD and UCLA) will be randomly selected to return approximately three months later to complete the same battery of assessments in the Behavioral and Neuroimaging Sessions to establish test-retest reliability of the latent constructs.

ELIGIBILITY:
1. Positive for anxiety and/or depressive symptoms.
2. Score on the PHQ-9 and OASIS.
3. Between the ages of 18-55, inclusive.
4. Have signed informed consent document(s) indicating that participant understands the purpose of and procedures required for the study and willing to participate in the study.
5. Have sufficient proficiency in English language to understand and complete interviews, questionnaires, and all other study procedures.
6. Have telephone or easy access to telephone.
7. History of brain injury with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study (to be determined by primary care provider).
8. Current and regular use of a medication that could affect brain functioning.
9. Must not have MRI contraindications such as: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a metal worker/welder, history of eye surgery/eyes washed out because of metal, inability to lie still on one's back for 60 minutes; prior neurosurgery; tattoos with metal dyes, unwillingness to remove body piercings, and pregnancy.
10. Intact or correctable vision and hearing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Investigators opted to identify individuals with anxiety or depression in a primary care setting, which investigators have used successfully to recruit a significant number of subjects, to maximize generalizability and external validity.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Relationship of latent constructs of positive and negative valence domains and neural indices of reward sensitivity and fear conditioning in treatment seeking depressed and anxious individuals. | 4 years
  Measure of BOLD % signal difference in brain regions of interest during reward or loss trials for anticipation and outcome phases in a reward paradigm, and conditioning trials in a fear conditioning paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Paulus, MD, Principal Investigator — UC San Diego; Murray B Stein, MD, MPH, Principal Investigator — UC San Diego
Locations (1):
- UCSD Psychiatry Clinical Research, La Jolla, California, United States

REFERENCES:
- [Background] Insel T, Cuthbert B, Garvey M, Heinssen R, Pine DS, Quinn K, Sanislow C, Wang P. Research domain criteria (RDoC): toward a new classification framework for research on mental disorders. Am J Psychiatry. 2010 Jul;167(7):748-51. doi: 10.1176/appi.ajp.2010.09091379. No abstract available. PMID 20595427
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Roy-Byrne P, Craske MG, Sullivan G, Rose RD, Edlund MJ, Lang AJ, Bystritsky A, Welch SS, Chavira DA, Golinelli D, Campbell-Sills L, Sherbourne CD, Stein MB. Delivery of evidence-based treatment for multiple anxiety disorders in primary care: a randomized controlled trial. JAMA. 2010 May 19;303(19):1921-8. doi: 10.1001/jama.2010.608. PMID 20483968

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03310398/Prot_SAP_000.pdf